CLINICAL TRIAL: NCT03527979
Title: Effect of Laparoscopic Ovarian Drilling on the Outcomes of in Vitro Fertilisation in Clomiphene-resistant Women With Polycystic Ovary Syndrome
Brief Title: Effect of Laparoscopic Ovarian Drilling on Outcomes of in Vitro Fertilisation in Clomiphene-resistant Women With Polycystic Ovary Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, rabab adel kamal, ob/gyn resident, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: rkamal
Record Dates: First submitted 2018-04-19; First posted 2018-05-17 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: PCOS

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCOS women with history of LOD before IVF/ICSI (Active Comparator)
  Interventions: Procedure: IVF/ICSI
- PCOS women without history of drilling (Active Comparator)
  Interventions: Procedure: IVF/ICSI

INTERVENTIONS:
Procedure: IVF/ICSI — IVF/ICSI

SUMMARY:
the polycystic ovarian syndrome is associated with an ovulation and infertility. recently the laparoscopic ovarian drilling has been used as surgical treatment for ovulation in women with polycystic ovarian syndrome, although its mechanism and outcomes are still unclear. this study is undertaken to evaluate the in vitro fertilisation outcomes in clomiphene-resistant women with PCOS who were treated with LOD.

ELIGIBILITY:
Inclusion Criteria:

* age between 25 and 35
* patients with established PCOS
* history at least one year infertility
* no response to clomiphene citrate for at least three cycles

Exclusion Criteria:

* history of previous IVF/ICSI
* chronic disease such as thyroid disorder and DM
* infertility due to sever male factor
* sever endometriosis
* infertility due to uterine factor such as multiple fibroid
* body mass index > 30

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate confirmed by b-hcg and visualizations of gestational sac by ultrasound | 3 months
  Pregnancy confirmed by b-hcg and visualization of gestational sac by ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university, Cairo, Egypt